CLINICAL TRIAL: NCT03783923
Title: A Multicenter Open-Label Study on the Safety and Efficacy of Deflazacort (Emflaza) in Subjects With Limb-Girdle Muscular Dystrophy 2I (LGMD2I)
Brief Title: A Study of Deflazacort (Emflaza®) in Participants With Limb-Girdle Muscular Dystrophy 2I (LGMD2I)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early due to low enrollment and missing efficacy assessment data due to missed visits related to COVID-19.
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCEMF-GD-004
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Results first posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-05

CONDITIONS: Limb-Girdle Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle | interventions — deflazacort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Deflazacort (Experimental): Participants will receive deflazacort 0.6 milligrams per kilograms per day (mg/kg/day) orally. The dose could be reduced in case of tolerability issues. Any participant assigned to placebo prior to the Version 4.0 amendment (prior to or after 01 February 2020) will have the option to be consented under Version 4.0 and will be switched to deflazacort for 26 weeks treatment. Any participant assigned to deflazacort prior to the Version 4.0 amendment (prior to 01 February 2020) will have the option to re-consent under Protocol Version 4.0 and continue for an additional 26 weeks treatment. Any participant assigned to deflazacort prior to the Version 4.0 amendment (after 01 February 2020) will have the option to re-consent under Protocol Version 4.0 at their Week 13 Visit and continue treatment until Week 26. Any new participant enrolled until 31 May 2020 will receive deflazacort for 26 weeks.
  Interventions: Drug: Deflazacort

INTERVENTIONS:
Drug: Deflazacort — Deflazacort tablet will be administered as per the dose and schedule specified in the arm.
  Other Names: Emflaza®

SUMMARY:
This study is designed to evaluate the safety and efficacy of deflazacort in participants with LGMD2I. Most participants enrolled will have a screening visit and 3 additional visits (after 1, 13, and 26 weeks of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of LGMD2I (confirmed mutation in the fukutin-related protein [FKRP] gene).
* Ability to ascend 4 stairs greater than or equal to (≥) 2.5 seconds and be able to complete the ascent and descent both at screening and baseline.
* Ability to understand the nature of the study and the consent form and to comply with study related procedures.
* Must weigh between 35 to 112.5 kilograms (kg).

Exclusion Criteria:

* Received ≥4 weeks of continuous, systemic corticosteroid therapy within 3 months of study screening visit.
* Presence of significant cardiomyopathy as defined by echocardiogram (left ventricular ejection fraction less than (<) 30 percent [%]) at screening.
* Requires fulltime ventilator support.
* History of chronic systemic fungal or viral infections.
* History of recent bacterial infection (including tuberculosis) per discretion of the Investigator.
* Diagnosis of diabetes mellitus (controlled and/or uncontrolled) defined as glycated hemoglobin (HbA1c) ≥6.5% (based on historical or present diagnosis).
* History of immunosuppression or other contraindications to glucocorticosteroid therapy.
* Requires concomitant use or greater than (>) 1 week of drugs or substances that are moderate to strong cytochrome P3A4 (CYP3A4) inhibitors (for example, clarithromycin, fluconazole, diltiazem, verapamil, grapefruit juice) or moderate or strong CYP3A4 inducers (that is, rifampin, efavirenz, carbamazepine, phenytoin) at baseline.
* Participated in an interventional clinical trial within the last 3 months prior the baseline visit.
* Unable or unwilling to comply with the contraceptive requirements of the protocol.
* Female participants who are pregnant and/or breastfeeding.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurologic, psychiatric, or allergic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristobal Passalacqua, MD, Study Director — PTC Therapeutics
Locations (18):
- United States (8):
  - Rare Disease Research, LLC, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Hugo W Moser Research Institute at Kennedy Krieger Institute, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Ottawa Hospital, Ottawa
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark
- France (2):
  - CHRU de NANCY Service de Neurologie, France
  - University Hospital La Timone, Marseille
- Ludwig-Maximilians University Munich, Friedrich-Baur-Institute, Munich, Germany
- Oslo University Hospital, Oslo, Norway
- Russia (2):
  - Pirogov Russian National Research Medical University, Moscow
  - Saint-Petersburg State Pediatric Medical University, Saint Petersburg
- Sahlgrenska University Hospital, Gothenburg, Sweden

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants enrolled under protocol v3.0 were 1:1 randomized to get placebo or deflazacort. After protocol v4.0, the study became an open-label study and all participants received deflazacort.
  Per planned analysis, participants who took at least 1 dose of deflazacort were pooled in the safety and efficacy summaries.
Groups:
- Deflazacort: Participants received deflazacort tablets, administered orally once daily at a target dose of 0.6 milligrams (mg)/kilograms (kg)/day for 26 weeks in placebo-controlled period and for 26 weeks in open-label extension period.
- Placebo: Participants received placebo matched to deflazacort tablets, administered orally once daily for 26 weeks in placebo-controlled period. Participants were then transitioned to receive deflazacort tablets, administered orally once daily at a target dose of 0.6 mg/kg/day for 26 weeks in open-label extension period.
Period: Placebo-Controlled Period (26 Weeks)
Arm/Group | Deflazacort | Placebo
Started | 5 | 6
Safety Population (Safety population included all enrolled participants who received at least 1 dose of deflazacort.) | 5 | 2 (2 participants who received placebo in placebo-controlled period transitioned to receive deflazacort in open-label extension.)
Completed (Open-label transition) | 1 | 2
Not Completed | 4 | 4
Not completed — Study Terminated | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Period: Open-Label Extension (26 Weeks)
Arm/Group | Deflazacort | Placebo
Started (Transited to Protocol V4 and Dosed under Open-Label) | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Study Terminated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled population included all informed-consented participants who met all inclusion and exclusion criteria.
Groups:
- Deflazacort: Participants received deflazacort tablets, administered orally once daily at a target dose of 0.6 mg/kg/day.
- Total: Total of all reporting groups
Arm/Group | Deflazacort | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Time to Climb 4 Stairs After 26 Weeks of Treatment With Deflazacort
Time Frame: Baseline, Week 26
Population: Safety population included all enrolled participants who received at least 1 dose of deflazacort. Here, 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Deflazacort
Number analyzed (Participants) | 7
seconds
  Baseline | 5.476 (2.0178)
  Change at Week 26: number analyzed (Participants) | 1
  Change at Week 26 | -0.200

2. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) After 26 Weeks of Treatment With Deflazacort
Time Frame: Baseline, Week 26
Population: Due to early termination of the study and missing efficacy assessment data due to missed visits related to COVID-19, data was not collected or analyzed for this secondary efficacy endpoint.
Arm/Group | Deflazacort
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in 2-Minute Walk Test After 26 Weeks of Treatment of Deflazacort
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Deflazacort
Number analyzed (Participants) | 7
meters
  Baseline | 135.4 (26.75)
  Change at Week 26: number analyzed (Participants) | 1
  Change at Week 26 | 2.0

4. Secondary Outcome: Change From Baseline in Time to up and go After 26 Weeks of Treatment With Deflazacort
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Deflazacort
Number analyzed (Participants) | 7
seconds
  Baseline | 11.93 (4.743)
  Change at Week 26: number analyzed (Participants) | 1
  Change at Week 26 | 9.70

5. Secondary Outcome: Change From Baseline in Time to Descend 4 Stairs After 26 Weeks of Treatment With Deflazacort
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Deflazacort
Number analyzed (Participants) | 7
seconds
  Baseline | 3.66 (1.707)
  Change at Week 26: number analyzed (Participants) | 1
  Change at Week 26 | 0.10

6. Secondary Outcome: Change From Baseline in Time to Run/Walk 10 Meters After 26 Weeks of Treatment With Deflazacort
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Deflazacort
Number analyzed (Participants) | 7
seconds
  Baseline | 8.53 (1.897)
  Change at Week 26: number analyzed (Participants) | 1
  Change at Week 26 | -0.40

7. Secondary Outcome: Change From Baseline in Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) After 26 Weeks of Treatment With Deflazacort
Time Frame: Baseline, Week 26
Population: as for outcome 2
Arm/Group | Deflazacort
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Hand-Held Myometry After 26 Weeks of Treatment With Deflazacort
Time Frame: Baseline, Week 26
Population: as for outcome 2
Arm/Group | Deflazacort
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline in Global T2 Relaxation Time of Selected Upper and Lower Limb Muscles After 26 Weeks of Treatment With Deflazacort
Time Frame: Baseline, Week 26
Population: as for outcome 2
Arm/Group | Deflazacort
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'. AEs were summarized separately for Stage 1 and for the overall ataluren experience.
Time Frame: Baseline up to Week 52
Population: Safety population included all enrolled participants who received at least 1 dose of deflazacort. Per planned analysis, participants who took at least 1 dose of deflazacort were pooled in the safety summaries. The participants who received only placebo during the study were not included for safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Deflazacort
Number analyzed (Participants) | 7
Participants | 5

11. Secondary Outcome: Area Under the Concentration Curve From Time Zero to t (AUC0-t) of 21-desacetyl Deflazacort and 6β-hydroxy-21-desacetyl Deflazacort
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose at Baseline and Week 13
Population: The pharmacokinetic (PK) population included all enrolled participants who received at least 1 dose of deflazacort and had at least one PK profile. Here, 'Number analyzed' = participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: nanograms (ng)*hour (hr)/milliliter (mL)
Arm/Group | Deflazacort
Number analyzed (Participants) | 4
nanograms (ng)*hour (hr)/milliliter (mL)
  21-desacetyl deflazacort: Baseline | 401.1 (139.62)
  21-desacetyl deflazacort: Week 13: number analyzed (Participants) | 2
  21-desacetyl deflazacort: Week 13 | 365.6 (NA) — Due to concentration below the limit of quantitation (BLQ) of 0.50 ng/mL, data not calculated.
  6β-hydroxy-21-desacetyl deflazacort: Week 1 | 418.2 (58.569)
  6β-hydroxy-21-desacetyl deflazacort: Week 13: number analyzed (Participants) | 2
  6β-hydroxy-21-desacetyl deflazacort: Week 13 | 515.3 (NA) — Due to concentration BLQ of 0.50 ng/mL, data not calculated.

12. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Infinity (AUC0-inf) of 21-desacetyl Deflazacort and 6β-hydroxy-21-desacetyl Deflazacort
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose at Baseline and Week 13
Population: The PK population included all enrolled participants who received at least 1 dose of deflazacort and had at least one PK profile. Here, 'Number analyzed' = participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Deflazacort
Number analyzed (Participants) | 4
ng*hr/mL
  21-desacetyl deflazacort: Baseline | 423.6 (150.16)
  21-desacetyl deflazacort: Week 13: number analyzed (Participants) | 0
  6β-hydroxy-21-desacetyl deflazacort: Week 1: number analyzed (Participants) | 3
  6β-hydroxy-21-desacetyl deflazacort: Week 1 | 520.3 (31.508)
  6β-hydroxy-21-desacetyl deflazacort: Week 13: number analyzed (Participants) | 0

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of 21-desacetyl Deflazacort and 6β-hydroxy-21-desacetyl Deflazacort
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose at Baseline and Week 13
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Deflazacort
Number analyzed (Participants) | 4
ng/mL
  21-desacetyl deflazacort: Baseline | 184.8 (49.054)
  21-desacetyl deflazacort: Week 13: number analyzed (Participants) | 2
  21-desacetyl deflazacort: Week 13 | 171.0 (NA) — Due to concentration BLQ of 0.50 ng/mL, data not calculated.
  6β-hydroxy-21-desacetyl deflazacort: Week 1 | 135.8 (29.205)
  6β-hydroxy-21-desacetyl deflazacort: Week 13: number analyzed (Participants) | 2
  6β-hydroxy-21-desacetyl deflazacort: Week 13 | 162.0 (NA) — Due to concentration BLQ of 0.50 ng/mL, data not calculated.

14. Secondary Outcome: Time to Reach Cmax (Tmax) of 21-desacetyl Deflazacort and 6β-hydroxy-21-desacetyl Deflazacort
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose at Baseline and Week 13
Population: as for outcome 12
Measure: Median (Full Range); unit: hr
Arm/Group | Deflazacort
Number analyzed (Participants) | 4
hr
  21-desacetyl deflazacort: Baseline | 0.992 [0.50 to 1.00]
  21-desacetyl deflazacort: Week 13: number analyzed (Participants) | 2
  21-desacetyl deflazacort: Week 13 | 0.525 [0.50 to 0.55]
  6β-hydroxy-21-desacetyl deflazacort: Week 1 | 1.000 [1.00 to 1.90]
  6β-hydroxy-21-desacetyl deflazacort: Week 13: number analyzed (Participants) | 2
  6β-hydroxy-21-desacetyl deflazacort: Week 13 | 1.550 [1.10 to 2.00]

15. Secondary Outcome: Half-Life (t1/2) of 21-desacetyl Deflazacort and 6β-hydroxy-21-desacetyl Deflazacort
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose at Baseline and Week 13
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Deflazacort
Number analyzed (Participants) | 4
hr
  21-desacetyl deflazacort: Baseline | 1.174 (0.0849)
  21-desacetyl deflazacort: Week 13: number analyzed (Participants) | 2
  21-desacetyl deflazacort: Week 13 | 1.235 (NA) — Due to concentration BLQ of 0.50 ng/mL, data not calculated.
  6β-hydroxy-21-desacetyl deflazacort: Week 1: number analyzed (Participants) | 3
  6β-hydroxy-21-desacetyl deflazacort: Week 1 | 2.358 (0.5825)
  6β-hydroxy-21-desacetyl deflazacort: Week 13: number analyzed (Participants) | 1
  6β-hydroxy-21-desacetyl deflazacort: Week 13 | 1.95

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: Safety population included all enrolled participants who received at least 1 dose of deflazacort. Per planned analysis, participants who took at least 1 dose of deflazacort were pooled in the safety summaries. The participants who received only placebo (not deflazacort) during the study were not monitored for safety assessments (including AE monitoring) per planned analysis.
Arm/Group | Deflazacort
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Deflazacort (N=7)
Cushingoid (Endocrine disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Influenza (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Weight increased (Investigations) | 2
Increased appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Visual field defect (Nervous system disorders) | 1
Apathy (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1/5 — This is a gender-specific AE. Only female participants were at risk.
Menstruation irregular (Reproductive system and breast disorders) | 1/5 — This is a gender-specific AE. Only female participants were at risk.
Acne (Skin and subcutaneous tissue disorders) | 2
Abnormal hair growth (Skin and subcutaneous tissue disorders) | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to low enrollment and missing efficacy assessment data due to missed visits related to COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT03783923/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT03783923/SAP_001.pdf